CLINICAL TRIAL: NCT03948906
Title: Comparing Post-stroke Functioning and Rehabilitation Pathways in a Region of North of Norway and a Region of Denmark. A Prospective Cohort Study.
Brief Title: Stroke and Rehabilitation in North of Norway and Central Denmark
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: Regionshospitalet Hammel Neurocenter (Other)
Responsible Party: Principal Investigator, Audny Anke, Professor, University Hospital of North Norway
Other Study IDs: SF 1175-14NCT02311426
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Stroke, Acute
Keywords: Stroke; Observational study; Rehabilitation; Health related quality of life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-stroke prospective multicenter cohort study. The objectives of the study was to compare functioning and health related quality of life in the two study regions, in relation to known predictors and to differences in organization of treatment- and rehabilitation. The inclusion was of consecutive acute stroke patients with ICD10 diagnosis I.63 and I.61 from a regional part of Northern Norway and Jylland Denmark. All were referred to stroke units. At baseline national stroke registry data were collected in each country. A questionnaire package was mailed to the participants 3- and 12-months post stroke. Telephone interviews at 3 months post stroke added information on functioning and rehabilitation.

DETAILED DESCRIPTION:
Post-stroke prospective multicenter cohort study. The objectives of the study was to compare functioning and health related quality of life in the two study regions, in relation to known predictors and to differences in organization of treatment- and rehabilitation. The inclusion was of consecutive acute stroke patients with ICD10 diagnosis I.63 and I.61 from a regional part of Northern Norway and Jylland Denmark. All were referred to stroke units. At baseline national stroke registry data were collected in each country. Telephone interviews at 3 months post stroke added information on functioning and rehabilitation. A questionnaire package was mailed to the participants 3- and 12-months post stroke. These included validated Questionnaires like QOLIBRI-OS, HADS, SS-QOL and EQ5D.

Validity studies on QOLIBRI-OS and SS-QOL has been published, along with several other papers. Synne Garder Pedersen and Guri Heiberg have finished their PhDs.

ELIGIBILITY:
* Clinical diagnosis acute ischemic or hemmorhagic stroke
* Inclusion period Mars 2014 to January 2016
* Hospitalised in Stroke Units
* Living in a defined geographic area in North of Norway or in Central Denmark

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ischemic or hemorrhagic stroke
Sampling Method: Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
HRQOL | 2014- 2016
  HRQOL measured by QOLIBRI-OS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pedersen SG, Heiberg GA, Nielsen JF, Friborg O, Stabel HH, Anke A, Arntzen C. Validity, reliability and Norwegian adaptation of the Stroke-Specific Quality of Life (SS-QOL) scale. SAGE Open Med. 2018 Jan 8;6:2050312117752031. doi: 10.1177/2050312117752031. eCollection 2018. PMID 29344360
- [Result] Heiberg G, Pedersen SG, Friborg O, Nielsen JF, Holm HS, Steinbuchel von N, Arntzen C, Anke A. Can the health related quality of life measure QOLIBRI- overall scale (OS) be of use after stroke? A validation study. BMC Neurol. 2018 Jul 18;18(1):98. doi: 10.1186/s12883-018-1101-9. PMID 30021558